CLINICAL TRIAL: NCT00000834
Title: A Phase I Study of Methotrexate for HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DATRI 013; 11742 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Methotrexate; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Lamivudine; Disease Progression; Anti-Inflammatory Agents; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Disease Progression | interventions — Lamivudine; Methotrexate; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Methotrexate
Drug: Zidovudine

SUMMARY:
To determine the safety and tolerance of methotrexate in HIV-infected patients. To determine the dose effective in modulating key markers of immune activation. To determine a dose suitable for Phase II or III evaluation in HIV-infected patients.

In HIV infection, complete immunological clearance of the foreign antigen does not occur, resulting in chronic immune activation. Because chronic immune activation may contribute to disease progression in HIV infection, immunomodulators may have therapeutic value in early HIV disease prior to development of opportunistic infections. The clinical benefits of methotrexate appear to derive from an anti-inflammatory effect; thus, it may reduce the state of chronic immune activation.

DETAILED DESCRIPTION:
In HIV infection, complete immunological clearance of the foreign antigen does not occur, resulting in chronic immune activation. Because chronic immune activation may contribute to disease progression in HIV infection, immunomodulators may have therapeutic value in early HIV disease prior to development of opportunistic infections. The clinical benefits of methotrexate appear to derive from an anti-inflammatory effect; thus, it may reduce the state of chronic immune activation.

Patients are randomized to receive methotrexate at Dose 1 or 2 (low doses) for 12 weeks, with 8 weeks of follow-up. If interim safety monitoring and viral burden results for the two cohorts support continuation, a third cohort of patients receive methotrexate starting at Dose 2 for the first 2 weeks, then at Dose 3 for the next 2 weeks, and at Dose 4 for the remaining 8 weeks, with 8 weeks of follow-up.

AS PER AMENDMENT 1/10/97:

The Dose 1 (the lowest dose) has been eliminated; the first 10 patients are now assigned to the next higher dose. Depending upon the results of interim safety data, the next cohort will be entered on the escalating dose regimen.

Also per this amendment, all patients will receive zidovudine and lamivudine for 30 days prior to the initiation of methotrexate, during the 12 weeks of methotrexate administration, and for the 8 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiemetics and antidiarrheals.
* Acetaminophen.
* Oral hypoglycemic agents.

PER AMENDMENT 5/15/96:

* Stable dose of antiretroviral (must be stable for at least 1 month prior to study entry). [AS

PER AMENDMENT 1/10/97:

* Combination zidovudine/lamivudine or zidovudine alone.]

Patients must have:

* HIV seropositivity.
* CD4 count >= 300 cells/mm3.
* No AIDS-defining condition.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptom or condition are excluded:

* Current positive PPD.

Concurrent Medication:

Excluded:

* Immunosuppressive or immunomodulatory drugs.
* Chronic nonsteroidal anti-inflammatory agents.
* Newly initiated antiretrovirals.
* Bone marrow suppressive drugs (e.g., TMP/SMX).

Concurrent Treatment:

AS PER AMENDMENT 1/10/97: Excluded:

* Antiretroviral therapy other than combination zidovudine/lamivudine or zidovudine alone; no initiation of other antiretroviral therapy should be planned while patient is on methotrexate.

Patients with the following prior conditions are excluded:

* Prior malignancies.
* Prior mucocutaneous herpes infection requiring antiviral therapy [AS PER AMENDMENT 7/31/96: Prior mucocutaneous herpes infection requiring systemic treatment with an antiviral agent (e.g., acyclovir); history of topical antiviral therapy is permitted].
* Anergic on DTH skin test within the past month (PER AMENDMENT 5/15/96: patients who are positive on DTH skin test but unable to receive the HIV-1 skin test because of allergies to insects, bee stings, etc., remain eligible for study enrollment).
* Inflammatory bowel disease, peptic ulcer disease, obesity combined with insulin-requiring diabetes, liver disease, or chronic renal disease within the past 6 months.
* Positive for HBsAg or hepatitis C antibody within the past 2 weeks.
* Chest radiograph within the past 60 days that shows cavity disease, infiltrates, or scars from prior disease that would preclude diagnosis of a new infectious process or drug-induced pneumonitis.

AS PER AMENDMENT 1/10/97:

* History of intolerance to zidovudine or lamivudine.

Prior Medication:

Excluded:

* Prior chemotherapy for malignancy.

Prior Treatment:

Excluded:

* Prior radiotherapy for malignancy. Alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egorin M, Study Chair; Fox L, Study Chair
Locations (7):
- United States (7):
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - New England Med Ctr, Boston, Massachusetts
  - Harper Hosp, Detroit, Michigan
  - Community Research Initiative on AIDS, New York, New York
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas